CLINICAL TRIAL: NCT05165745
Title: Stick2PrEP Women/Trans Individuals: Increasing Pre-Exposure Prophylaxis (PrEP) Uptake, Adherence, and Retention in Care, and Understanding PrEP Preferences Among Predominantly Black and Latinx Cisgender Women and Transgender Individuals
Brief Title: Stick2PrEP Cisgender Women and Trans Individuals
Acronym: S2P:CWTI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Magdalena Sobieszczyk, Harold C. Neu Professor of Infectious Diseases (in Medicine) at the Columbia University Medical Center, Columbia University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: AAAS6460
Record Dates: First submitted 2021-12-08; First posted 2021-12-21 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: HIV Prevention; Pre-exposure Prophylaxis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Cisgender Women and Trans Individuals (CWTI) (Other): Cisgender women and trans individuals (CWTI) who are taking PrEP, have considered and decided not to take PrEP, or who have discontinued PrEP.
  Interventions: Behavioral: Individualized Feedback

INTERVENTIONS:
Behavioral: Individualized Feedback — Participants taking PrEP will receive questionnaires regarding self-reported weekly PrEP adherence; they will then receive individualized text-message or email feedback based on their self-reported adherence.

SUMMARY:
Taking a daily anti-HIV pill can protect people from HIV infection. This is called preexposure prophylaxis [PrEP]. Many cisgender women and trans individuals do not know this medication is available; others struggle to take the pill every day. It is important to understand attitudes and preferences about HIV prevention options, especially as new options become available. This study plans to evaluate preferences over time among cisgender women and trans individuals who are taking medication to prevent HIV, and among cisgender women and trans individuals who are not taking medication but are at risk of HIV. The investigators enroll up to 175 participants who visit the HIV prevention clinic, and the investigators will ask participants to complete questionnaires at regular follow up visits and between visits. This study may help the investigators understand how best to prevent HIV among people at risk.

DETAILED DESCRIPTION:
Participants will receive online questionnaires about demographic characteristics, social determinants of health, and preferences regarding PrEP modalities. Qualitative, in-depth surveys will be conducted with 12 CWTI who decide not to start PrEP and 12 CWTI who decide to discontinue PrEP to explore the drivers behind those decisions. Participants who are taking PrEP will be offered the option of providing dried blood spot samples at clinic visits to measure PrEP levels and will receive an online questionnaire addressing their preferences regarding different modalities of measuring PrEP levels. The purpose of the HemaSpot™ kit is to understand the subjects' perceptions of using this kit for self-testing PrEP levels; this will inform future strategies regarding PrEP monitoring. Participants taking PrEP will also receive questionnaires regarding self-reported weekly PrEP adherence; they will then receive individualized text-message or email feedback based on their self-reported adherence in addition to standard-of-care retention/adherence counseling. Participants on PrEP can also elect to receive or emails messages to remind them to take PrEP and attend follow up appointments.

ELIGIBILITY:
Inclusion Criteria:

* Cisgender women and trans individuals who have an indication for PrEP and have 1) decided to take PrEP, 2) decided not to take PrEP, or 3) decided to discontinue PrEP

Exclusion Criteria:

* Cannot provide informed consent
* Living with HIV

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Cisgender women and transgender individuals
Enrollment: 175 (Estimated)
Dates: Start 2021-10-25 (Actual); Primary Completion 2026-10-25 (Estimated); Study Completion 2026-10-25 (Estimated)

PRIMARY OUTCOMES:
Correlation Between PrEP modality preference and PrEP initiation/persistence in care | 12 months
  Description of CWTI's preferences for different PrEP modalities and the relationship between preference and PrEP initiation/persistence in care. Preferences are evaluated using questionnaires developed by the study team; questions include ranked choice and Likert score responses. Persistence in care is measured by using the electronic medical record to track sexual health care visits over study period.
PrEP Measurement Preferences Scale Score | 12 months
  CWTI's experience with and preferences regarding laboratory measurement techniques for PrEP. Preferences are evaluated based on a questionnaire developed by the study team; acceptability, feasibility, and perceived usefulness of varying PrEP measurement techniques are evaluated using a 5-point Likert scale. Scores range from 0 to 5, with a higher score indicating greater acceptability, feasibility, and usefulness.
Percentage of participants on PrEP who remain engaged in sexual health care | 12 months
  Effect of individualized feedback on retention in care at 12 months. Retention in care is measured by using the electronic medical record to track sexual health care visits over the study period. Outcome will be measured by percentage of participants on PrEP who remain engaged in sexual health care (attending visits) at study center through 12 months after enrollment.

SECONDARY OUTCOMES:
Correlation of risk factors for low PrEP adherence and retention | 12 months
  Risk factors that may be associated with poor retention in PrEP/sexual health care and low adherence to PrEP. Adherence to PrEP is measured by weekly self-report among participants taking PrEP. Retention in sexual healthcare is measured by review of the electronic medical record to track sexual health care visits over the study period.
Web-Based App User Satisfaction Score | 12 months
  User comfort/satisfaction with the web-based app will be assessed using Likert scale responses. Scores range from 0 to 5 with a higher score indicating greater user comfort/satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: Magdalena Sobieszczyk, MD, MPH, Principal Investigator — Columbia University
Locations (1):
- Columbia University Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No